CLINICAL TRIAL: NCT01642355
Title: Investigation of Motivational Interviewing and Prevention Consults to Achieve Cardiovascular Targets
Brief Title: Prevention Trial to Achieve Cardiovascular Targets
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: The Rainer Arnhold Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMPACT-2012-400
Record Dates: First submitted 2012-07-03; First posted 2012-07-17 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Disease; Peripheral Arterial Disease; Hyperlipidemia; Hypertension; Diabetes; Prediabetes; Obesity
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Hyperlipidemias; Hypertension; Diabetes Mellitus; Prediabetic State; Obesity | interventions — Referral and Consultation; Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (No Intervention): Usual care includes physician assistant and/or nurse based medical and lifestyle recommendations in consultation with cardiac catheterization attending or patient's clinical cardiologist to potentially improve the patient's medical and lifestyle regimen. Relevant educational material is routinely distributed to patients.
- Prevention Consult (Active Comparator): In addition to usual care, patients will receive a prevention consult by a prevention fellow and attending following their intervention. The consult will include guideline based medical recommendations for optimization of the patient's medical regimen targeting dyslipidemia, hypertension and diabetes. In addition, each patient will be educated on the cardiovascular disease process and given detailed lifestyle recommendations on physical activity, improved nutrition, smoking cessation and medication adherence.
  Interventions: Behavioral: Prevention Consult
- Consult & Behavioral Intervention (Active Comparator): In addition to usual care and prevention consult (as detailed above), patients will receive a full motivational intervention program by a trained motivational coach and text messages over 6 months.
  Interventions: Behavioral: Consult & Behavioral Intervention

INTERVENTIONS:
Behavioral: Prevention Consult — In addition to usual care, patients will receive a prevention consult by a prevention fellow and attending following their intervention. The consult will include guideline based medical recommendations for optimization of the patient's medical regimen targeting dyslipidemia, hypertension and diabetes. In addition, each patient will be educated on the cardiovascular disease process and given detailed lifestyle recommendations on physical activity, improved nutrition, smoking cessation and medication adherence.
  Arms: Prevention Consult
Behavioral: Consult & Behavioral Intervention — In addition to usual care and prevention consult (as detailed above), patients will receive a full motivational intervention program by a trained motivational coach and text messages over 6 months.
  Arms: Consult & Behavioral Intervention

SUMMARY:
The objective of IMPACT (Investigation of Motivational Interviewing and Prevention Consults to Achieve Cardiovascular Targets) is to determine the best management strategy for patients undergoing cardiovascular intervention. IMPACT is a prospective randomized trial that will enroll 400 patients post-cardiovascular intervention. The study will compare different cardiovascular prevention strategies: (1) usual care, (2) cardiovascular prevention consult, and (3) cardiovascular prevention consult with a behavioral intervention program over a 6-month period. The trial hypothesis is that for patients undergoing a cardiovascular intervention, a prevention consult and behavioral intervention is superior to usual care in reducing cardiovascular risk. The primary endpoint will be non-HDL cholesterol. Secondary endpoints include other lipid values, metabolic risk, smoking cessation, physical activity, nutritional status, medication adherence and quality of life. IMPACT is scheduled to begin enrollment in the June of 2012.

DETAILED DESCRIPTION:
SPECIFIC AIMS

Primary aim:

The primary aim is that a targeted Cardiovascular Prevention consult will reduce non-HDL cholesterol compared to usual care at 6 months post-intervention.

Secondary aim:

The secondary aim is that a targeted Cardiovascular Prevention consult plus a behavioral intervention will reduce non-HDL cholesterol compared to usual care at 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* at least 21 years of age or older
* Subjects scheduled to undergo a percutaneous coronary or peripheral vascular intervention
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Life expectancy less than 1-year
* Inability to walk

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2012-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reduction of Non-HDL cholesterol | 6 months

SECONDARY OUTCOMES:
Lipids | 6 months
  LDL-C, HDL, triglycerides
Metabolic risk factors | 6 months
  weight, BMI, HbA1C, abdominal circumference
Physical Activity | 6 months
  Yale Physical Activity assessment (Part 2)
Nutrition | 6 months
  Northwest Lipid Research Clinic (NWLRC) Fat Intake Score and fruit and vegetable assessment questions
Medication Adherence | 6 months
  Morisky-4 medication adherence survey
Optimal medical regimen | 6 months
  assessment of lipid lowering and cardiovascular medication regimen
Quality of life | 6 months
  Euro Qual 5D survey
Smoking cessation | 6 months
  Patient-based Assessment and Counseling for Physical Activity and Nutrition (PACE) smoking assessment
Cardiovascular risk | 6 months
  cardiovascular risk assessment score (i.e. Framingham)
Cardiovascular events | 5 years
  cardiovascular events and hospitalizations reported by phone call follow-up up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Gianos, M.D., Principal Investigator — NYU Langone Health; Jeffrey S Berger, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

REFERENCES:
- [Background] Gianos E, Schoenthaler A, Mushailov M, Fisher EA, Berger JS. Rationale and design of the Investigation of Motivational Interviewing and Prevention Consults to Achieve Cardiovascular Targets (IMPACT) trial. Am Heart J. 2015 Sep;170(3):430-7.e9. doi: 10.1016/j.ahj.2015.06.001. Epub 2015 Jun 6. PMID 26385025
- [Derived] Gianos E, Schoenthaler A, Guo Y, Zhong J, Weintraub H, Schwartzbard A, Underberg J, Schloss M, Newman JD, Heffron S, Fisher EA, Berger JS. Investigation of Motivational Interviewing and Prevention Consults to Achieve Cardiovascular Targets (IMPACT) trial. Am Heart J. 2018 May;199:37-43. doi: 10.1016/j.ahj.2017.12.019. Epub 2018 Jan 9. PMID 29754664
- See also: New York University Langone Center for the Prevention of Cardiovascular Disease website — http://www.med.nyu.edu/cvprevention/